CLINICAL TRIAL: NCT00577668
Title: UARK 2007-01, A Phase II Pilot Study of the Combination of Melphalan, Bortezomib, Thalidomide and Dexamethasone (MEL-VTD) and Autologous Transplantation for Patients Relapsing or Progressing After Tandem Transplantation
Brief Title: A Pilot Study of the Combination of Melphalan, Bortezomib, Thalidomide and Dexamethasone (MEL-VTD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Mauricio Pineda-Roman, MD, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-01
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Bortezomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VDT and Melphalan (Experimental): To find out if three drugs, bortezomib, thalidomide, and dexamethasone in addition to high doses of melphalan (M-VTD) and autologous transplant can be given safely and effectively to subjects who have failed previous regimens with transplant(s).
  Interventions: Drug: Melphalan, Velcade, Thalidomide, Dexamethasone

INTERVENTIONS:
Drug: Melphalan, Velcade, Thalidomide, Dexamethasone — To assess, in patients with one or two prior auto transplants, the efficacy of a high-dose combination chemotherapy with MEL 300 (in 3 fractions of 100 mg/m2 on days -7, -4, -1) plus VTD (Velcade = bortezomib 1.3 mg/m2 on days -7, -4, -1; Thalidomide 200 mg/d on days -1 through -7; Dexamethasone 40 mg on days -7, -6, -4, -3, -1, 0) followed by autologous peripheral blood stem cell (PBSC) infusion of a minimum dose of 3 million CD34 cells/kg.

SUMMARY:
In this study, researchers want to find out if using the VTD regimen, along with higher doses melphalan, in subjects who have relapsed or progressed after previous transplant(s), can be given safely to subjects who have failed previous transplant(s).

DETAILED DESCRIPTION:
Autologous transplant is now considered a standard treatment for many patients with multiple myeloma. An autologous transplant is a procedure in which stem cells are removed from a patient and then given back to the patient following intensive treatment. Doctors remove healthy stem cells from a patient's circulating blood system and store them before the patient receives high-dose chemotherapy. The stem cells are then returned to the patient, where they can produce new blood cells to replace cells destroyed by the treatment. The drug usually used before transplant is melphalan alone in 1 or 2 high doses. In past studies conducted at UAMS, researchers have shown that a chemotherapy treatment regimen called "VTD" is effective in patients with multiple myeloma who have failed previous treatments. VTD is a combination of drugs consisting of VelcadeTM (also known as bortezomib), Thalidomide, and Dexamethasone. In this study, researchers want to find out if using the VTD regimen, along with higher doses melphalan, in subjects who have relapsed or progressed after previous transplant(s) can be given safely to subjects who have failed previous transplant(s).

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented MM with relapsed or progressive disease after either scheduled tandem or one autologous transplantation.
* Patient has measurable disease in which to capture response.
* Performance status of 2 as per Zubroid scale, unless PS of 3-4 based solely on bone pain.
* Patients must have a platelet count 75,000/μL, and an ANC of at least 1,000/μL.
* Patients must have adequate renal function defined as serum creatinine < 2.5 mg/dL.
* Patients must have adequate hepatic function defined as serum transaminases and direct bilirubin < 2 x the upper limit of normal.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Male or female adults of at least 18 years of age.
* Patients must have signed an IRB-approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations.

Exclusion Criteria:

* Chemotherapy or radiotherapy received within the previous 2 weeks.
* Significant neurotoxicity, defined as grade > 2 neurotoxicity per NCI Common Toxicity Criteria (See Appendix).
* Platelet count < 75,000/mm3, or ANC < 1,000/μl.
* Clinically significant hepatic dysfunction as noted by bilirubin or AST > 3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association (NYHA) Class III or Class IV heart failure.
* Myocardial infarction within the last 6 months.
* Uncontrolled, active infection requiring IV antibiotics.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly controlled hypertension, diabetes mellitus, or other serious or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Pregnant or potential for pregnancy. Women of childbearing potential will have a pregnancy test at screening, and will be required to use a medically approved contraceptive method.
* Breast-feeding women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
VTD regimen with melphalan | 12 months
  To find out if using the VTD regimen, along with higher doses melphalan, in subjects who have relapsed or progressed after previous transplant(s), can be given safely to subjects who have failed previous transplant(s).

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Pineda-Roman, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States